CLINICAL TRIAL: NCT02795247
Title: Three Dimensional Computed Tomography Comparison of the Transtibial, Modified Transtibial and Anteromedial Portal Technique for Recreation of the Anterior Cruciate Ligament Anatomic Footprint
Brief Title: Comparison of 3 Techniques for Recreation of Anterior Cruciate Ligament Anatomic Footprint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OrthoCarolina Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPORT037
Record Dates: First submitted 2016-06-06; First posted 2016-06-10 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Anterior Cruciate Ligament Reconstruction
MeSH Terms: interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hybrid Transtibial Technique (Active Comparator): Reconstruction of the ACL using the hybrid transtibial technique
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Accessory Anteromedial Portal Technique (Active Comparator): Reconstruction of the ACL using the accessory anteromedial portal technique
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction
- Transtibial Technique (Active Comparator): Reconstruction of the ACL using the transtibial technique.
  Interventions: Procedure: Anterior Cruciate Ligament Reconstruction

INTERVENTIONS:
Procedure: Anterior Cruciate Ligament Reconstruction
  Other Names: ACL Reconstruction

SUMMARY:
The purpose of this study is to compare the tomographic results of patients who underwent single-bundle anterior cruciate ligament reconstruction at the investigator's institution using the transtibial, accessory medial portal technique and the modified transtibial technique to determine which technique best recreates the anterior cruciate ligament anatomic footprint.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for single bundle ACL reconstruction, with or without associated partial meniscectomy or meniscal repair.
* Skeletally mature patients
* Patients who are able and willing to receive post-operative CT imaging of the affected knee

Exclusion Criteria:

* Previous ACL reconstruction in the studied knee
* Previous ACL injury or reconstruction in the contralateral kneeConcomitant non-ACL ligament reconstruction or osteotomy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-26 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
3D reconstructed CT imaging | 6 weeks Post-Operatively
  Used to measure tunnel position.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | 6 weeks post-operative
  Change in IKDC subjective knee evaluation since before surgery
Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks post-operative
  Change in KOOS since before surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | 6 months post-operative
  Change in IKDC subjective knee evaluation since before surgery
Knee injury and Osteoarthritis Outcome Score (KOOS) | 6 months post-operative
  Change in KOOS since before surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | 1 year post-operative
  Change in IKDC subjective knee evaluation since before surgery
Knee injury and Osteoarthritis Outcome Score (KOOS) | 1 year post-operative
  Change in KOOS since before surgery
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation | 2 year post-operative
  Change in IKDC subjective knee evaluation since before surgery
Knee injury and Osteoarthritis Outcome Score (KOOS) | 2 year post-operative
  Change in KOOS since before surgery
Knee Laxity | 6 month post-operatively
  Pivot shift test will be used to a measure of knee laxity

CONTACTS AND LOCATIONS:
Overall Officials: Dana P Piasecki, MD, Principal Investigator — OrthoCarolina Research Institute, Inc.
Locations (1):
- OrthoCarolina Sports Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robin BN, Jani SS, Marvil SC, Reid JB, Schillhammer CK, Lubowitz JH. Advantages and Disadvantages of Transtibial, Anteromedial Portal, and Outside-In Femoral Tunnel Drilling in Single-Bundle Anterior Cruciate Ligament Reconstruction: A Systematic Review. Arthroscopy. 2015 Jul;31(7):1412-7. doi: 10.1016/j.arthro.2015.01.018. Epub 2015 Mar 5. PMID 25749530
- [Background] Youm YS, Cho SD, Eo J, Lee KJ, Jung KH, Cha JR. 3D CT analysis of femoral and tibial tunnel positions after modified transtibial single bundle ACL reconstruction with varus and internal rotation of the tibia. Knee. 2013 Aug;20(4):272-6. doi: 10.1016/j.knee.2012.10.024. Epub 2012 Nov 26. PMID 23195998
- [Background] Lee MC, Seong SC, Lee S, Chang CB, Park YK, Jo H, Kim CH. Vertical femoral tunnel placement results in rotational knee laxity after anterior cruciate ligament reconstruction. Arthroscopy. 2007 Jul;23(7):771-8. doi: 10.1016/j.arthro.2007.04.016. PMID 17637414
- [Background] Alentorn-Geli E, Lajara F, Samitier G, Cugat R. The transtibial versus the anteromedial portal technique in the arthroscopic bone-patellar tendon-bone anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2010 Aug;18(8):1013-37. doi: 10.1007/s00167-009-0964-0. Epub 2009 Nov 10. PMID 19902178
- [Background] Takeda Y, Iwame T, Takasago T, Kondo K, Goto T, Fujii K, Naruse A. Comparison of tunnel orientation between transtibial and anteromedial portal techniques for anatomic double-bundle anterior cruciate ligament reconstruction using 3-dimensional computed tomography. Arthroscopy. 2013 Feb;29(2):195-204. doi: 10.1016/j.arthro.2012.08.020. Epub 2012 Dec 24. PMID 23270788
- [Background] de Abreu-e-Silva GM, de Oliveira MH, Maranhao GS, Deligne Lde M, Pfeilsticker RM, Novais EN, Nunes TA, de Andrade MA. Three-dimensional computed tomography evaluation of anterior cruciate ligament footprint for anatomic single-bundle reconstruction. Knee Surg Sports Traumatol Arthrosc. 2015 Mar;23(3):770-6. doi: 10.1007/s00167-013-2703-9. Epub 2013 Oct 22. PMID 24146049
- [Background] Larson AI, Bullock DP, Pevny T. Comparison of 4 femoral tunnel drilling techniques in anterior cruciate ligament reconstruction. Arthroscopy. 2012 Jul;28(7):972-9. doi: 10.1016/j.arthro.2011.12.015. Epub 2012 Mar 10. PMID 22409948
- [Background] Osaki K, Okazaki K, Matsubara H, Kuwashima U, Murakami K, Iwamoto Y. Asymmetry in Femoral Tunnel Socket Length During Anterior Cruciate Ligament Reconstruction With Transportal, Outside-In, and Modified Transtibial Techniques. Arthroscopy. 2015 Dec;31(12):2365-70. doi: 10.1016/j.arthro.2015.06.026. Epub 2015 Aug 24. PMID 26315055
- [Background] Bernard M, Hertel P, Hornung H, Cierpinski T. Femoral insertion of the ACL. Radiographic quadrant method. Am J Knee Surg. 1997 Winter;10(1):14-21; discussion 21-2. PMID 9051173
- [Background] Forsythe B, Kopf S, Wong AK, Martins CA, Anderst W, Tashman S, Fu FH. The location of femoral and tibial tunnels in anatomic double-bundle anterior cruciate ligament reconstruction analyzed by three-dimensional computed tomography models. J Bone Joint Surg Am. 2010 Jun;92(6):1418-26. doi: 10.2106/JBJS.I.00654. PMID 20516317
- [Background] Sohn OJ, Lee DC, Park KH, Ahn HS. Comparison of the Modified Transtibial Technique, Anteromedial Portal Technique and Outside-in Technique in ACL Reconstruction. Knee Surg Relat Res. 2014 Dec;26(4):241-8. doi: 10.5792/ksrr.2014.26.4.241. Epub 2014 Dec 2. PMID 25505707
- [Derived] Trofa DP, Saltzman BM, Corpus KT, Connor PM, Fleischli JE, Piasecki DP. A Hybrid Transtibial Technique Combines the Advantages of Anteromedial Portal and Transtibial Approaches: A Prospective Randomized Controlled Trial. Am J Sports Med. 2020 Nov;48(13):3200-3207. doi: 10.1177/0363546520956645. Epub 2020 Oct 5. PMID 33017169